CLINICAL TRIAL: NCT00537576
Title: A Phase I Study of the Safety of LACTIN-V Administered Vaginally to Healthy Women
Brief Title: Safety Study of Lactobacillus Administered Vaginally to Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Osel, Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: LV-005
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2014-04

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Low dose LACTIN-V applicator (Experimental): Low dose LACTIN-V applicator (150 mg LACTIN-V, 5.0 x 10^8 CFU), administered vaginally once a day for 5 consecutive days
  Interventions: Biological: Low dose LACTIN-V applicator
- Medium dose LACTIN-V applicator (Experimental): Medium dose LACTIN-V applicator (300 mg LACTIN-V, 1.0 x 10^9 CFU), administered vaginally once a day for 5 consecutive days
  Interventions: Biological: Medium dose LACTIN-V applicator
- High dose LACTIN-V applicator (Experimental): High dose LACTIN-V applicator (600 mg LACTIN-V, 2.0 x 10^9 CFU), administered vaginally once a day for 5 consecutive days
  Interventions: Biological: High dose LACTIN-V applicator
- Low dose Placebo applicator (Placebo Comparator): Low dose Placebo applicator (150 mg Placebo), administered vaginally once a day for 5 consecutive days
  Interventions: Other: Low dose Placebo applicator
- Medium dose Placebo applicator (Placebo Comparator): Medium dose Placebo applicator (300 mg Placebo), administered vaginally once a day for 5 consecutive days
  Interventions: Other: Medium dose Placebo
- High dose Placebo applicator (Placebo Comparator): High dose Placebo applicator (600 mg Placebo), administered vaginally once a day for 5 consecutive days
  Interventions: Other: High dose Placebo applicator

INTERVENTIONS:
Biological: Low dose LACTIN-V applicator — Low dose LACTIN-V applicator (150 mg LACTIN-V, 5.0 x 10^8 CFU), administered vaginally once a day for 5 consecutive days
  Other Names: Lactobacillus crispatus CTV-05
  Arms: Low dose LACTIN-V applicator
Biological: Medium dose LACTIN-V applicator — Medium dose LACTIN-V applicator (300 mg LACTIN-V, 1.0 x 10^9 CFU), administered vaginally once a day for 5 consecutive days
  Other Names: Lactobacillus crispatus CTV-05
  Arms: Medium dose LACTIN-V applicator
Biological: High dose LACTIN-V applicator — High dose LACTIN-V applicator (600 mg LACTIN-V, 2.0 x 10^9 CFU), administered vaginally once a day for 5 consecutive days
  Other Names: Lactobacillus crispatus CTV-05
  Arms: High dose LACTIN-V applicator
Other: Low dose Placebo applicator — Low dose Placebo applicator (150 mg Placebo), administered vaginally once a day for 5 consecutive days
  Other Names: Control substance
  Arms: Low dose Placebo applicator
Other: Medium dose Placebo — Medium dose Placebo applicator (300 mg Placebo), administered vaginally once a day for 5 consecutive days
  Other Names: Control substance
  Arms: Medium dose Placebo applicator
Other: High dose Placebo applicator — High dose Placebo applicator (600 mg Placebo), administered vaginally once a day for 5 consecutive days
  Other Names: Control substance
  Arms: High dose Placebo applicator

SUMMARY:
The purpose of this study is to compare the safety, tolerability, and acceptability of LACTIN-V (Active Ingredient: Lactobacillus crispatus CTV-05) with a matching placebo at three doses using pre-filled vaginal applicators in healthy pre-menopausal women. The study hypothesis is that LACTIN-V will be safe, tolerable, and acceptable at each dose and will not differ significantly from the placebo controls.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate that LACTIN-V is safe, well tolerated, and acceptable to healthy pre-menopausal women when administered vaginally using pre-filled applicators at doses of 150 mg (5.0 x 10^8 CFU), 300 mg (1.0 x 10^9 CFU), or 600 mg (2.0 x 10^9 CFU) daily for 5 consecutive days as compared to placebo applicators containing 150 mg, 300 mg, or 600 mg of a matching placebo formulation without Lactobacillus crispatus CTV-05.

Safety will be assessed by:

* Incidence and severity of adverse events through assessing symptoms, physical examination findings, and signs of irritation involving the external genitalia, cervix or vagina, including disruption of the epithelium and blood vessels as seen on pelvic examination and colposcopy.
* Laboratory parameters including urinalysis, a complete blood count (CBC) with differential, and chemistry panels to assess systemic effects of the study product.

Tolerability will be assessed by:

* The proportion of participants who discontinue study product use due to overt adverse events
* The proportion of participants who complete the full dosing schedule

Acceptability will be assessed by:

- Self-administered questionnaires and focus group discussions about acceptability of the study product

ELIGIBILITY:
Inclusion Criteria:

* Healthy pre-menopausal women 18- 40 years of age at date of screening.
* Regular menstrual cycles (21-35 days) or amenorrheic for at least 3 months (long acting progestin contraceptives).
* Normal Pap smear collected at the screening visit.
* Previous sexual experience including vaginal intercourse.
* Previous experience of gynecological examinations.
* Currently in a mutually monogamous sexual relationship or not sexually active.
* Agree to be sexually abstinent thoughout the trial.
* Agree to abstain from the use of any other intravaginal product thoughout the trial
* Agree to use an adequate method of birth control for the duration of the study to avoid pregnancy.

Exclusion Criteria:

* Urogenital infection at screening or within the 21 days prior to screening (UTI, bacterial vaginosis, Trichomonas vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis, Treponema pallidum or Herpes simplex).
* History of recurrent genital herpes.
* Diagnosis of N. gonorrhoeae, C. trachomatis, T. pallidum or T. vaginalis on two or more occasions during the six months prior to screening.
* Pregnancy or within 2 months of last pregnancy.
* Lactation.
* Antibiotic or antifungal therapy within 30 days of enrollment visit.
* Concurrent investigational drug use within 30 days or 10 half-lives of the drug, of enrollment visit or during the study.
* Menopause.
* IUD insertion or removal, pelvic surgery, cervical cryotherapy or cervical laser within the last 3 months.
* Use of a NuvaRing® within 3 days of the screening visit or during the course of the study.
* New (less than 3 months)long-acting treatments (e.g. depot formulation including medroxyprogesterone acetate (DMPA) form of hormonal birth control). - - Diabetes or other significant disease or acute illness.
* Known HIV infection or positive HIV test at screening.
* Immunosuppressive drug within 60 days.
* Previous participation in a L. crispatus CTV-05 clinical study.
* Colposcopic findings at the enrollment visit involving significant deep disruption of the epithelium.
* Abnormal results for the pap smear at the screening visit.
* Known allergy to any component of LACTIN-V, other significant drug allergy or to latex (condoms).
* Known drug or alcohol abuse.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Cohen, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Giorgi A, Torriani S, Dellaglio F, Bo G, Stola E, Bernuzzi L. Identification of vaginal lactobacilli from asymptomatic women. Microbiologica. 1987 Oct;10(4):377-84. PMID 3695985
- [Background] Antonio MA, Hawes SE, Hillier SL. The identification of vaginal Lactobacillus species and the demographic and microbiologic characteristics of women colonized by these species. J Infect Dis. 1999 Dec;180(6):1950-6. doi: 10.1086/315109. PMID 10558952
- [Background] Antonio MA, Hillier SL. DNA fingerprinting of Lactobacillus crispatus strain CTV-05 by repetitive element sequence-based PCR analysis in a pilot study of vaginal colonization. J Clin Microbiol. 2003 May;41(5):1881-7. doi: 10.1128/JCM.41.5.1881-1887.2003. PMID 12734221
- [Background] Sobel JD. Vaginitis in adult women. Obstet Gynecol Clin North Am. 1990 Dec;17(4):851-79. PMID 2092246
- [Background] Thomason JL, Gelbart SM, Scaglione NJ. Bacterial vaginosis: current review with indications for asymptomatic therapy. Am J Obstet Gynecol. 1991 Oct;165(4 Pt 2):1210-7. doi: 10.1016/s0002-9378(12)90729-2. PMID 1951577
- [Background] Pastore LM, Thorp JM Jr, Royce RA, Savitz DA, Jackson TP. Risk score for antenatal bacterial vaginosis: BV PIN points. J Perinatol. 2002 Mar;22(2):125-32. doi: 10.1038/sj.jp.7210654. PMID 11896517
- [Background] Gibney L, Macaluso M, Kirk K, Hassan MS, Schwebke J, Vermund SH, Choudhury P. Prevalence of infectious diseases in Bangladeshi women living adjacent to a truck stand: HIV/STD/hepatitis/genital tract infections. Sex Transm Infect. 2001 Oct;77(5):344-50. doi: 10.1136/sti.77.5.344. PMID 11588280
- [Background] Kamara P, Hylton-Kong T, Brathwaite A, Del Rosario GR, Kristensen S, Patrick N, Weiss H, Figueroa PJ, Vermund SH, Jolly PE. Vaginal infections in pregnant women in Jamaica: prevalence and risk factors. Int J STD AIDS. 2000 Aug;11(8):516-20. doi: 10.1258/0956462001916425. PMID 10990336
- [Background] Goldenberg RL, Klebanoff MA, Nugent R, Krohn MA, Hillier S, Andrews WW. Bacterial colonization of the vagina during pregnancy in four ethnic groups. Vaginal Infections and Prematurity Study Group. Am J Obstet Gynecol. 1996 May;174(5):1618-21. doi: 10.1016/s0002-9378(96)70617-8. PMID 9065140
- [Background] Sewankambo N, Gray RH, Wawer MJ, Paxton L, McNaim D, Wabwire-Mangen F, Serwadda D, Li C, Kiwanuka N, Hillier SL, Rabe L, Gaydos CA, Quinn TC, Konde-Lule J. HIV-1 infection associated with abnormal vaginal flora morphology and bacterial vaginosis. Lancet. 1997 Aug 23;350(9077):546-50. doi: 10.1016/s0140-6736(97)01063-5. PMID 9284776
- [Background] Jurney TH, de Ruyter H, Vigersky RA. Cushing's disease presenting as amenorrhoea with hyperprolactinaemia: report of two cases. Clin Endocrinol (Oxf). 1981 Jun;14(6):539-45. doi: 10.1111/j.1365-2265.1981.tb02963.x. PMID 7197596
- [Background] Hay PE, Lamont RF, Taylor-Robinson D, Morgan DJ, Ison C, Pearson J. Abnormal bacterial colonisation of the genital tract and subsequent preterm delivery and late miscarriage. BMJ. 1994 Jan 29;308(6924):295-8. doi: 10.1136/bmj.308.6924.295. PMID 8124116
- [Background] Eschenbach DA. Bacterial vaginosis and anaerobes in obstetric-gynecologic infection. Clin Infect Dis. 1993 Jun;16 Suppl 4:S282-7. doi: 10.1093/clinids/16.supplement_4.s282. PMID 8324132
- [Background] Hawes SE, Hillier SL, Benedetti J, Stevens CE, Koutsky LA, Wolner-Hanssen P, Holmes KK. Hydrogen peroxide-producing lactobacilli and acquisition of vaginal infections. J Infect Dis. 1996 Nov;174(5):1058-63. doi: 10.1093/infdis/174.5.1058. PMID 8896509
- [Background] Puapermpoonsiri S, Kato N, Watanabe K, Ueno K, Chongsomchai C, Lumbiganon P. Vaginal microflora associated with bacterial vaginosis in Japanese and Thai pregnant women. Clin Infect Dis. 1996 Oct;23(4):748-52. doi: 10.1093/clinids/23.4.748. PMID 8909838
- [Background] Reid G, Burton J. Use of Lactobacillus to prevent infection by pathogenic bacteria. Microbes Infect. 2002 Mar;4(3):319-24. doi: 10.1016/s1286-4579(02)01544-7. PMID 11909742
- [Background] Hillier SL, Krohn MA, Klebanoff SJ, Eschenbach DA. The relationship of hydrogen peroxide-producing lactobacilli to bacterial vaginosis and genital microflora in pregnant women. Obstet Gynecol. 1992 Mar;79(3):369-73. doi: 10.1097/00006250-199203000-00008. PMID 1738516
- [Background] Avonts D, Sercu M, Heyerick P, Vandermeeren I, Meheus A, Piot P. Incidence of uncomplicated genital infections in women using oral contraception or an intrauterine device: a prospective study. Sex Transm Dis. 1990 Jan-Mar;17(1):23-9. PMID 2305333
- [Background] Soper DE, Bump RC, Hurt WG. Bacterial vaginosis and trichomoniasis vaginitis are risk factors for cuff cellulitis after abdominal hysterectomy. Am J Obstet Gynecol. 1990 Sep;163(3):1016-21; discussion 1021-3. doi: 10.1016/0002-9378(90)91115-s. PMID 2403128
- [Background] Workowski KA, Berman SM. CDC sexually transmitted diseases treatment guidelines. Clin Infect Dis. 2002 Oct 15;35(Suppl 2):S135-7. doi: 10.1086/342100. No abstract available. PMID 12353199
- [Background] Bukusi EA, Cohen CR, Meier AS, Waiyaki PG, Nguti R, Njeri JN, Holmes KK. Bacterial vaginosis: risk factors among Kenyan women and their male partners. Sex Transm Dis. 2006 Jun;33(6):361-7. doi: 10.1097/01.olq.0000200551.07573.df. PMID 16547451
- [Background] Eschenbach DA, Hillier S, Critchlow C, Stevens C, DeRouen T, Holmes KK. Diagnosis and clinical manifestations of bacterial vaginosis. Am J Obstet Gynecol. 1988 Apr;158(4):819-28. doi: 10.1016/0002-9378(88)90078-6. PMID 3259075
- [Background] Hillier SL, Kiviat NB, Hawes SE, Hasselquist MB, Hanssen PW, Eschenbach DA, Holmes KK. Role of bacterial vaginosis-associated microorganisms in endometritis. Am J Obstet Gynecol. 1996 Aug;175(2):435-41. doi: 10.1016/s0002-9378(96)70158-8. PMID 8765265
- [Background] Larsson PG, Platz-Christensen JJ, Thejls H, Forsum U, Pahlson C. Incidence of pelvic inflammatory disease after first-trimester legal abortion in women with bacterial vaginosis after treatment with metronidazole: a double-blind, randomized study. Am J Obstet Gynecol. 1992 Jan;166(1 Pt 1):100-3. doi: 10.1016/0002-9378(92)91838-2. PMID 1733176
- [Background] Eschenbach DA. Bacterial vaginosis: emphasis on upper genital tract complications. Obstet Gynecol Clin North Am. 1989 Sep;16(3):593-610. PMID 2687747
- [Background] Watts DH, Krohn MA, Hillier SL, Eschenbach DA. Bacterial vaginosis as a risk factor for post-cesarean endometritis. Obstet Gynecol. 1990 Jan;75(1):52-8. PMID 2296423
- [Background] Newton ER, Prihoda TJ, Gibbs RS. A clinical and microbiologic analysis of risk factors for puerperal endometritis. Obstet Gynecol. 1990 Mar;75(3 Pt 1):402-6. PMID 2406660
- [Background] Paavonen J, Teisala K, Heinonen PK, Aine R, Laine S, Lehtinen M, Miettinen A, Punnonen R, Gronroos P. Microbiological and histopathological findings in acute pelvic inflammatory disease. Br J Obstet Gynaecol. 1987 May;94(5):454-60. doi: 10.1111/j.1471-0528.1987.tb03125.x. PMID 3580330
- [Background] Larsson PG, Platz-Christensen JJ, Forsum U, Pahlson C. Clue cells in predicting infections after abdominal hysterectomy. Obstet Gynecol. 1991 Mar;77(3):450-2. PMID 1992415
- [Background] Kurki T, Sivonen A, Renkonen OV, Savia E, Ylikorkala O. Bacterial vaginosis in early pregnancy and pregnancy outcome. Obstet Gynecol. 1992 Aug;80(2):173-7. PMID 1635726
- [Background] Riduan JM, Hillier SL, Utomo B, Wiknjosastro G, Linnan M, Kandun N. Bacterial vaginosis and prematurity in Indonesia: association in early and late pregnancy. Am J Obstet Gynecol. 1993 Jul;169(1):175-8. doi: 10.1016/0002-9378(93)90157-e. PMID 8333449
- [Background] Hillier SL, Nugent RP, Eschenbach DA, Krohn MA, Gibbs RS, Martin DH, Cotch MF, Edelman R, Pastorek JG 2nd, Rao AV, et al. Association between bacterial vaginosis and preterm delivery of a low-birth-weight infant. The Vaginal Infections and Prematurity Study Group. N Engl J Med. 1995 Dec 28;333(26):1737-42. doi: 10.1056/NEJM199512283332604. PMID 7491137
- [Background] Silver HM, Sperling RS, St Clair PJ, Gibbs RS. Evidence relating bacterial vaginosis to intraamniotic infection. Am J Obstet Gynecol. 1989 Sep;161(3):808-12. doi: 10.1016/0002-9378(89)90406-7. PMID 2782365
- [Background] Hillier SL, Martius J, Krohn M, Kiviat N, Holmes KK, Eschenbach DA. A case-control study of chorioamnionic infection and histologic chorioamnionitis in prematurity. N Engl J Med. 1988 Oct 13;319(15):972-8. doi: 10.1056/NEJM198810133191503. PMID 3262199
- [Background] Taha TE, Hoover DR, Dallabetta GA, Kumwenda NI, Mtimavalye LA, Yang LP, Liomba GN, Broadhead RL, Chiphangwi JD, Miotti PG. Bacterial vaginosis and disturbances of vaginal flora: association with increased acquisition of HIV. AIDS. 1998 Sep 10;12(13):1699-706. doi: 10.1097/00002030-199813000-00019. PMID 9764791
- [Background] Martin HL, Richardson BA, Nyange PM, Lavreys L, Hillier SL, Chohan B, Mandaliya K, Ndinya-Achola JO, Bwayo J, Kreiss J. Vaginal lactobacilli, microbial flora, and risk of human immunodeficiency virus type 1 and sexually transmitted disease acquisition. J Infect Dis. 1999 Dec;180(6):1863-8. doi: 10.1086/315127. PMID 10558942
- [Background] Myer L, Denny L, Telerant R, Souza Md, Wright TC Jr, Kuhn L. Bacterial vaginosis and susceptibility to HIV infection in South African women: a nested case-control study. J Infect Dis. 2005 Oct 15;192(8):1372-80. doi: 10.1086/462427. Epub 2005 Sep 9. PMID 16170754
- [Background] Hay P. Recurrent Bacterial Vaginosis. Curr Infect Dis Rep. 2000 Dec;2(6):506-512. doi: 10.1007/s11908-000-0053-5. PMID 11095900
- [Background] Bradshaw CS, Morton AN, Hocking J, Garland SM, Morris MB, Moss LM, Horvath LB, Kuzevska I, Fairley CK. High recurrence rates of bacterial vaginosis over the course of 12 months after oral metronidazole therapy and factors associated with recurrence. J Infect Dis. 2006 Jun 1;193(11):1478-86. doi: 10.1086/503780. Epub 2006 Apr 26. PMID 16652274
- [Background] Myer L, Kuhn L, Denny L, Wright TC Jr. Recurrence of symptomatic bacterial vaginosis 12 months after oral metronidazole therapy in HIV-positive and -negative women. J Infect Dis. 2006 Dec 15;194(12):1797-9. doi: 10.1086/509625. No abstract available. PMID 17109360
- [Background] Hughes VL, Hillier SL. Microbiologic characteristics of Lactobacillus products used for colonization of the vagina. Obstet Gynecol. 1990 Feb;75(2):244-8. PMID 2300352
- [Background] Chimura T, Funayama T, Murayama K, Numazaki M. [Ecological treatment of bacterial vaginosis]. Jpn J Antibiot. 1995 Mar;48(3):432-6. Japanese. PMID 7752457
- See also: Click here for more information about this study: LACTIN-V phase I study — http://www.oselinc.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2007 and January 2008, 12 participants were recruited through advertising in health centers, educational institutions, community bulletin boards and online forums.
Pre-assignment Details: All 12 enrolled participants completed the study.
Groups:
- Low Dose Applicator: Low dose LACTIN-V applicator (150 mg LACTIN-V, 5.0 x 10^8 CFU) and Placebo applicator (150 mg Placebo), randomized 3:1
- Medium Dose Applicator: Medium dose LACTIN-V applicator (300 mg LACTIN-V, 1.0 x 10^9 CFU) and Placebo applicator (300 mg), randomized 3:1
- High Dose Applicator: High dose LACTIN-V applicator (600 mg LACTIN-V, 2.0 x 10^9 CFU) and Placebo applicator (600 mg Placebo), randomized 3:1
- Placebo Control Substance Low Dose: Placebo control substance Low Dose contained a nutrient matrix of 150 mg per dose.
- Placebo Control Substance Medium Dose: Placebo control substance Medium Dose contained a nutrient matrix of 300 mg per dose.
- Placebo Control Substance High Dose: Placebo control substance High Dose contained a nutrient matrix of 600 mg per dose.
Period: Overall Study
Arm/Group | Low Dose Applicator | Medium Dose Applicator | High Dose Applicator | Placebo Control Substance Low Dose | Placebo Control Substance Medium Dose | Placebo Control Substance High Dose
Started | 3 | 3 | 3 | 1 | 1 | 1
Completed | 3 | 3 | 3 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Applicator | Medium Dose Applicator | High Dose Applicator | Placebo Control Substance Low Dose | Placebo Control Substance Medium Dose | Placebo Control Substance High Dose | Total
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 1 | 1 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 1 | 1 | 1 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (7.0) | 29.1 (7) | 29.1 (7.0) | 29.1 (7) | 29.1 (7) | 29.1 (7) | 29.1 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 1 | 1 | 1 | 12
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 1 | 1 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety of LACTIN-V in Healthy Pre-menopausal Women.
Description: Safety was measured by comparing the number of women experiencing adverse events of grade 3 or higher during the study.
Time Frame: 35 days
Population: The analysis was per protocol. Number of participants for descriptive analysis only.
Measure: Number; unit: participants
Arm/Group | Low Dose Applicator | Medium Dose Applicator | High Dose Applicator | Placebo Control Substance Low Dose | Placebo Control Substance Medium Dose | Placebo Control Substance High Dose
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 1 | 1
participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Tolerability of LACTIN-V in a Pre-filled Applicator.
Description: Tolerability was measured as proportion of women remaining in the study, and NOT prematurely exiting the trial due to an adverse event.
Time Frame: 35 days
Population: Analysis per Protocol. Number of participants for descriptive analysis.
Measure: Number; unit: participants
Arm/Group | Low Dose Applicator | Medium Dose Applicator | High Dose Applicator | Placebo Control Substance Low Dose | Placebo Control Substance Medium Dose | Placebo Control Substance High Dose
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 1 | 1
participants | 3 | 3 | 3 | 1 | 1 | 1

3. Secondary Outcome: Acceptability of LACTIN-V in Pre-filled Applicators
Description: Acceptability and overall satisfaction with the study product was measured using the response to the following question: "I would use the product again" with the following response options (strongly agree, agree, neutral, disagree, strongly disagree)
  Acceptability is reported as the number of women in each group who strongly agreed or agreed with the statement that they would use the product again.
Time Frame: 35 days
Measure: Number; unit: participants
Arm/Group | Low Dose Applicator | Medium Dose Applicator | High Dose Applicator | Placebo Control Substance Low Dose | Placebo Control Substance Medium Dose | Placebo Control Substance High Dose
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 1 | 1
participants | 3 | 3 | 2 | 1 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Low Dose Applicator | Medium Dose Applicator | High Dose Applicator | Placebo Control Substance Low Dose | Placebo Control Substance Medium Dose | Placebo Control Substance High Dose
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 1/1 | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Applicator (N=3) | Medium Dose Applicator (N=3) | High Dose Applicator (N=3) | Placebo Control Substance Low Dose (N=1) | Placebo Control Substance Medium Dose (N=1) | Placebo Control Substance High Dose (N=1)
vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — expected AE
Abdominal pain (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
headache (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vaginal odor (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
vaginal candidiasis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No